CLINICAL TRIAL: NCT06290804
Title: Evaluation of Educational Activity for Increasing Environmentally Sustainable Behaviors and Awareness of Climate Change Health Effects in 60-72 Month Old Children
Brief Title: Assessing Sustainable Behaviors and Health Impacts of Climate Change
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ezgi Yucel, research asistant, medical doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: drezgiyucel0000000193593877
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Climate Change; Child Health
Keywords: Climate Change; Sustainability; Impacts of Climate Change on Child Health
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children aged 60-72 months-before (Other): As a data collection tool, two separate questionnaires were prepared for parents and children by utilizing the literature. The questionnaire form prepared for children consists of 3 parts. The first part includes some variables thought to be related to climate change and sustainability, the second part includes the questions '' Environmental Sustainability Scale for 60-72 Month-old Children" and the third part includes questions about health effects of climate change.
  The questionnaire form prepared before the intervention will be applied to children who agree to participate in the study.
  Interventions: Other: education
- Children aged 60-72 months-after (Other): In the intervention phase, the effectiveness of the training program and training videos to be applied to children will be evaluated in terms of sustainable behaviors towards the environment and awareness of the health effects of climate change in 60-72 month old children.
  Interventions: Other: education

INTERVENTIONS:
Other: education — Training program on Health Impacts of Sustainable Behaviors and Climate Change

SUMMARY:
The relationship between climate change, sustainability and child health is complex and important. These three concepts are interacting factors and have significant impacts on children's health. Sustainability measures are vital to protect child health by mitigating the impacts of climate change. At the same time, children's education and awareness is an important factor that will contribute to future generations living in a sustainable world. As a society, tackling climate change and striving for a sustainable future is crucial to ensure that children live healthy and safe lives. The aim of this study is to evaluate the effectiveness of the education program and educational videos to be applied to children in terms of environmentally sustainable behaviors and awareness of the health effects of climate change in 60-72-month-old children studying in Eskişehir Odunpazarı Municipality Day Care Center and Nurseries. In addition, in this study, it was aimed to measure the level of global climate change awareness of parents and to evaluate the relationship with children's environmentally sustainable behaviors.

DETAILED DESCRIPTION:
The data will be obtained from 60-72 month old children and their parents who are studying in Day Care Centers and Nurseries of Eskişehir Odunpazarı Municipality in 2023-2024.

Within the scope of the study, a detailed explanation of the study, informed consent forms and questionnaire forms will be delivered to the parents and children through their teachers. The questionnaire form prepared by utilizing the literature will be applied to the parents and children who agree to participate in the study. Subsequently, the education program to be prepared for the intervention group will be implemented in selected day care centers and nurseries. Four weeks after the educational intervention, the children will be reached again and the children in the intervention group will be asked to fill out the questionnaire form for the second time.

The population of the study consisted of 132 children aged 60-72 months who were studying in Day Care Centers and Nurseries of Eskişehir Odunpazarı Municipality in 2023-2024.

In the study, when type 1 (α) error was taken as 5% and type 2 error (1-β) was taken as 90%, it was calculated with the G*Power 3.1 statistical program that there should be at least 36 people in the intervention group when the effect size was accepted as 0.50. Considering those who could not continue the study, it was planned to be conducted with a total of 38 students in order to reach the required sample size.

ELIGIBILITY:
Inclusion Criteria:

* The study will include children aged 60-72 months and their parents, whose consent was obtained from parents and children.

Exclusion Criteria:

* Children with any condition that prevents them from attending school (any chronic medical condition that prevents them from participating in the study) and mainstreaming students (children in need of special education; children with adaptation difficulties, dyslexia, autism diagnosis, attention deficit and hyperactivity disorder) will not be included in the study.

Ages: 60 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
increasing sustainable behaviors | 6 months
  Changes in the ''Environmental Sustainability Scale for 60-72 Months Old'' score. The questionnaire form prepared for children consists of 3 parts. The first section includes some variables that are thought to be related to climate change and sustainability, and the second section includes '' Environmental Sustainability Scale for 60-72 Month-old Children" and the third part includes questions about the health effects of climate change.
raising awareness of the health impacts of climate change | 6 months
  Changes in the total score for questions on the effects of climate change on children's health.
raising awareness of global climate change | 6 months
  As a data collection tool, two separate questionnaires were prepared for parents and children by utilizing the literature. The parent questionnaire consists of three parts. The first part includes sociodemographic characteristics of parents and children (age of the parent, age of the child (month), gender of the parent, gender of the child, parental education level, occupation of the parent, family income status), the second part includes some variables thought to be related to climate change awareness, sustainability and health effects of climate change, and the third part includes the questions of the "Global Climate Change Awareness Scale".

CONTACTS AND LOCATIONS:
Locations (1):
- Ezgi Yücel, Odunpazari, Eskişehir, Turkey (Türkiye)